CLINICAL TRIAL: NCT04307420
Title: Postoperative Pain Following Restoration With Sonic Fill Versus Composite Resin in Children With Deep Carious First Permanent Molar: A Randomized Clinical Pilot Study
Brief Title: Postoperative Pain Following Restoration With Composite Resin Versus Sonic Fill
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mennatallah Samy Mohamed Maklad, Principle Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Composite Resin VS Sonic Fill
Record Dates: First submitted 2020-03-11; First posted 2020-03-13 (Actual); Last update posted 2020-07-16 (Actual); Status verified 2020-07

CONDITIONS: Postoperative Pain
Keywords: First Permanent Molar; Composite; Sonic Fill; Resin Restoration; Pediatric Dentistry
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sonic Fill Restoration (Experimental): Using sonic activation system turns the highly filled sonic fill composite into a flowable which enables the material to rapidly fill the cavity effortlessly- greatly reducing procedure time.
  Interventions: Procedure: Sonic Fill Restoration
- Composite Resin Restoration (Active Comparator): Direct composite restorations are the most requested and performed dental procedures. The incremental placement technique is the gold standard for posterior universal composite placement.
  Interventions: Procedure: Composite Resin Restoration

INTERVENTIONS:
Procedure: Sonic Fill Restoration — Kerr's Sonic Fill is the only sonic-activated, single-step, bulk-fill composite that starts out as a low-viscosity composite.
  Arms: Sonic Fill Restoration
Procedure: Composite Resin Restoration — Composite resins are polymer-based materials used in dentistry for aesthetic repairs.Polymerization is accomplished typically with a hand held curing light that emits specific wavelengths keyed to the initiator and catalyst packages involved.
  Arms: Composite Resin Restoration

SUMMARY:
The aim of this study is to assess the postoperative pain following restoration with composite resin versus sonic fill in children with deep carious first permanent molar.

DETAILED DESCRIPTION:
For many years, composite resin restorations have been considered an acceptable treatment choice for anterior applications. Recent advances in composite resin mechanical properties and improved adhesive systems have broadened the application of these materials to include the restoration of posterior teeth. However, it is still generally accepted that posterior composite resin restorations have limitations and that there is no ideal material available. A volumetric shrinkage occurs when a composite resin material is cured. The shrinkage is the result of conversion of monomer molecules into a more dense polymer network, which leads to bulk contraction. A new nanohybrid composite activated by sonic energy has been recently introduced as a single-step, bulk-fill restorative material. This system utilizes the patented sonic-activation technology enabling a rapid flow of composite into the cavity for effortless placement and superior adaptation in one single layer, thereby, emphasizes its practical and efficient technique for placing posterior composites. The hand piece, designed by KaVo (Germany), delivers sonic energy at varying intensities, which is adjusted on the shank from low to high (1 to 5) to control rate of composite extrusion.

ELIGIBILITY:
Inclusion Criteria:

* Asymptomatic First Permanent Molar
* Age of the patient ranging from 6-9 years
* Normal periodontal status
* Teeth with no previous restorative treatment
* Good oral health
* Absences of pathological mobility

Exclusion Criteria:

* Adverse medical history
* Potential behavioral problems
* Parents refusing participation of their children

Ages: 6 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 32 (Estimated)
Dates: Start 2020-09-01 (Estimated); Primary Completion 2021-05-31 (Estimated); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative Pain | Baseline
  The primary outcome (postoperative pain) is evaluated the following day of the treatment performed by a phone call from the outcome assessor, a week and a month after to check in any pain.

SECONDARY OUTCOMES:
Clinical Evaluation of Restoration (Modified USPHS Criteria) | 3 months, 6 months, 9 months
  The secondary outcome (USPHS) is evaluated by the outcome assessor and an investigator using the given scores as follows: The modified United States Public Health Service (USPHS) criteria for retention, color matching, marginal discoloration, marginal adaptation, secondary caries, surface texture and anatomical form were used.

CONTACTS AND LOCATIONS:
Overall Officials: Nevine Waly, Profesor, Study Director — Cairo University

REFERENCES:
- [Background] Chandrasekhar V, Rudrapati L, Badami V, Tummala M. Incremental techniques in direct composite restoration. J Conserv Dent. 2017 Nov-Dec;20(6):386-391. doi: 10.4103/JCD.JCD_157_16. PMID 29430088
- [Background] Afifi SMH, Haridy MF, Farid MR. Evaluation of Post-Operative Sensitivity of Bulk Fill Resin Composite versus Nano Resin Composite: A Randomized Controlled Clinical Study. Open Access Maced J Med Sci. 2019 Jul 26;7(14):2335-2342. doi: 10.3889/oamjms.2019.656. eCollection 2019 Jul 30. PMID 31592052
- [Result] Atabek D, Aktas N, Sakaryali D, Bani M. Two-year clinical performance of sonic-resin placement system in posterior restorations. Quintessence Int. 2017;48(9):743-751. doi: 10.3290/j.qi.a38855. PMID 28849804